CLINICAL TRIAL: NCT00347256
Title: Preoperative Radiotherapy and Concomitant Chemotherapy Followed by Surgery for Advanced Paranasal Sinus Carcinoma
Brief Title: Chemoradiotherapy Followed by Surgery for Advanced Paranasal Sinus Cancer
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tennessee (Other)
Collaborators: North American Skull Base Society (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NASBS-PNS001
Record Dates: First submitted 2006-06-29; First posted 2006-07-04 (Estimated); Last update posted 2008-12-10 (Estimated); Status verified 2008-12

CONDITIONS: Paranasal Sinus Neoplasms
MeSH Terms: conditions — Paranasal Sinus Neoplasms | interventions — Cisplatin; Radiotherapy; Transurethral Resection of Bladder

INTERVENTIONS:
Drug: cisplatin
Procedure: targeted radiation therapy
Procedure: tumor resection

SUMMARY:
The purpose of this study is to determine the efficacy of concurrent chemotherapy and radiotherapy pre-operatively in patients with advanced paranasal sinus cancer. The main objectives of this study are: 1) to measure the rate of complete response to preoperative chemoradiation and 2) to study the efficacy of combining preoperative chemoradiation and surgery in terms of local control of the cancer two years post treatment.

ELIGIBILITY:
Inclusion Criteria:

* Karnofsky Performance Score: >= 60
* Creatinin clearance >= 50 ml/min or serum creatinine =<1.5 mg/dl
* Total bilirubin, AST, ALT =< 1.5 X laboratory uln
* ANC >= 2000/mm3, platelets >= 100,000/mm3
* Serum calcium within normal range
* T3 or T4 state tumors of paranasal sinuses
* Squamous cell carcinoma, adenocarcinoma, high-grade mucoepidermoid carcinoma, sinonasal undifferentiated carcinoma

Exclusion Criteria:

* History of other malignancy in the last 3 years
* Other serious comorbidity that may significantly reduce the survival in next 5 years
* Pregnant or lactating women
* History of radiation to the head and neck region
* Paranasal sinus tumor is recurrent after prior treatment
* Presence of cervical node metastasis
* Presence of distant metastasis
* Advanced nasopharyngeal malignancy with sphenoid or posterior ethmoid invasion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)

PRIMARY OUTCOMES:
Local control of cancer at two years post treatment
Response to preoperative chemoradiation

SECONDARY OUTCOMES:
Estimation of the proportion of the inoperable tumors which become operable after chemoradiation
Identification of factors that are associated with inoperability
Estimation of the overall survival and cumulative incidence of death due to disease at 2 years
Determination of the acute and long-term toxicity, particularly ophthalmologic complications, and surgical morbidity associated with this regimen
Measurement of the accuracy of conventional imaging techniques (CT, MRI) compared with the addition of PET imaging in predicting the response to chemoradiation therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Sandeep Samant, MS, FRCS, Study Chair — University of Tennessee; Sandeep Samant, MS, FRCS, Principal Investigator — University of Tennessee

REFERENCES:
- See also: North American Skull Base Society webpage — http://www.nasbs.org